CLINICAL TRIAL: NCT04256434
Title: A Bioavailability Study of NALDEBAIN ER Injection and Nalbuphine Injection in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LT1001-104
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Health
MeSH Terms: interventions — sebacoyl dinalbuphine ester; Nalbuphine

STUDY DESIGN:
Intervention Model Description: This is an open-label, sequential 2 cohort, intramuscular injection study in healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dinabuphine sebacate (Experimental): Each subject in cohort 1 will receive 150 mg Dinalbuphine sebacate (75 mg/mL x 2 mL) intramuscularly.
  Interventions: Drug: Dinalbuphine sebacate
- Nalbuphine HCl (Active Comparator): Each subject in cohort 2 will receive 20 mg Nalbuphine (20 mg x 1 mL) intramuscularly.
  Interventions: Drug: Nalbuphine HCl

INTERVENTIONS:
Drug: Dinalbuphine sebacate — 150 mg Dinalbuphine sebacate
  Other Names: NALDEBAIN ER Injection; Sebacoyl Dinalbuphine Ester Injection; LT1001
  Arms: Dinabuphine sebacate
Drug: Nalbuphine HCl — 20 mg Nalbuphine
  Other Names: Nalbuphine HCl Injection
  Arms: Nalbuphine HCl

SUMMARY:
This is an open-label, sequential 2 cohort, intramuscular injection study in healthy volunteers. The study will enroll approximately 24 healthy volunteers to examine the safety, pharmacokinetics, and bioavailability after intramuscular injection of NALDEBAIN ER Injection and nalbuphine injection.

DETAILED DESCRIPTION:
Each subject in a cohort will be evaluated for study eligibility during the screening period, which is within 28 days prior to receiving the study drug (Day 1). Eligible subjects will be admitted into the study site on Day -1 and will be required to stay in clinical site for 5 (Cohort 1) or 2 nights (Cohort 2) for study procedures in each cohort. Eligible subjects will undergo additional eligibility assessments on Day -1 and those reconfirmed eligible will intramuscularly receive NALDEBAIN ER Injection (Cohort 1) or nalbuphine (Cohort 2) on Day 1.

The blood sampling timepoints for Cohort 1 will be at predose, 6, 12, 24, 48, 56, 64, 72, 80, 88, and 96 hours after dosing. Subjects will be discharged after the 96-hour blood sample and return to the clinical site for the sample collection at 120, 168, 216, 288 and 360 hours post dosing. The blood sampling timepoints for Cohort 2 will be predose, 5, 15, and 30 minutes postdose, and 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose.

Subjects will return for a follow-up visit to complete safety evaluations for approximately 15 days after study drug administration in cohort 1; and 1 days after study drug administration in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 55 years of age inclusive at the time of signing the informed consent form
2. Body weight must be above 60 kg.
3. Body Mass Index (BMI) 18 to 40 kg/m2
4. In good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
5. If male, must agree to use contraception as detailed in Appendix 5 of this protocol during the treatment period until the final PK sample, and refrain from donating sperm for 90 days after the dosing.
6. If female, is not pregnant (see Appendix 5), not breastfeeding, and at least one of the following conditions applies:

   Not a woman of childbearing potential (WOCBP) as defined in Appendix 5 OR A WOCBP who agrees to follow the contraceptive guidance in Appendix 5 during the treatment period until the last PK sample.
7. Vital signs (after 3 minutes resting in a semi-supine position) which are within the following ranges:

   * Oral temperature between 35.0-37.5°C.
   * Systolic blood pressure, 90-140 mm Hg.
   * Diastolic blood pressure, 50-90 mm Hg.
   * Pulse rate, 50-90 bpm.
   * Respiratory rate, 12-20 bpm
   * Oxyhemoglobin saturation, ≥95%
8. Fasting blood glucose, <110 mg/dL.
9. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. Use of any prescription medications or over-the-counter, non-prescription preparations (including herbal preparations) within 2 weeks prior to study entry unless deemed acceptable by the Investigator (except up to 5 doses of ≤ 1000 mg of acetaminophen or ≤ 400 mg ibuprofen within this 2 weeks period).
2. Alcohol or caffeine ingested within 72 hours prior to dosing.
3. Significant illness within 2 weeks prior to dosing.
4. Participation in any clinical investigation within 2 months prior to dosing or longer as required by local regulation.
5. Donation or loss of more than 500 mL of blood within 3 months prior to dosing. Donation or loss of more than 250 mL of blood within 2 months prior to dosing.
6. Documented history of cardiovascular disease.
7. Documented history of gastrointestinal disease.
8. Documented history of asthma or lung disease.
9. Presence of liver disease or liver injury as indicated by an abnormal liver function profile such as aspartate aminotransaminase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (gamma-GT), Alkaline Phosphatase, or Total Bilirubin at Screening. (value of AST or ALT above 3 times of the upper limit of the normal range; other items clinically significant abnormality judged by investigator).
10. Presence of impaired renal function as indicated by abnormal creatinine or BUN values or abnormal urinary constituents at Screening. (value of creatinine or BUN beyond the range from -20% of the lower limit of the normal range to +20% of the upper limit of the normal range; other items clinically significant abnormality judged by investigator)
11. Documented history of neurological disease.
12. Documented history of psychiatric disease.
13. Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or tests positive for HBsAg or anti-HCV at Screening.
14. A known hypersensitivity to nalbuphine or its analogs.
15. History of drug or alcohol abuse within 12 months prior to dosing or positive test results for alcohol or drugs of abuse at Screening and admission.
16. Permanent confinement to an institution.
17. Pregnant or lactating women.
18. Subject has received any investigational product within 30 days or 5 half-lives (whichever is longer) prior to the dosing day or is planning to participate in a clinical trial during the study period.
19. Has preplanned surgery or procedures that would interfere with the conduct of the study
20. Individuals are judged by the investigator to be undesirable subjects for other reasons.
21. Is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Bioavailability of nalbuphine after intramuscular injection of NALDEBAIN and Nalbuphine. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  To evaluate the relative bioavailability of nalbuphine after intramuscular injection of NALDEBAIN and Nalbuphine.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  Cmax for NALDEBAIN and Nalbuphine.
Tmax of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  Tmax for NALDEBAIN and Nalbuphine.
AUCinf of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  AUCinf for NALDEBAIN and Nalbuphine.
AUClast of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  AUClast for NALDEBAIN and Nalbuphine.
Elimination half-life (t1/2) of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  Elimination half-life for NALDEBAIN and Nalbuphine.
Total body clearance of the drug from plasma (CL) of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  Total body clearance for NALDEBAIN and Nalbuphine.
Volume of distribution (Vd) of nalbuphine, sebacoyl mononalbuphine ester (SME) and dinalbuphine sebacate. | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  Volume of distribution for NALDEBAIN and Nalbuphine.
Incidence and severity of adverse events (AEs) | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  To evaluate the systemic and local safety and tolerance.
Number of subjects with AEs | Cohort 1: From predose to 360 hours post dosing. Cohort 2 : From predose to 24 hours post dosing.
  To evaluate number of subjects with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: David Nguyen, MD, Principal Investigator — WCCT Global
Locations (1):
- WCCT Global Inc., Cypress, California, United States